Title: The practice of providing palliative care in the situation of the COVID-19 pandemic in the perspective of physicians and nurses – survey study (PEOpLe-C19 study)

## **Authors:**

Tereza Prokopova M.D.<sup>1</sup>
Jan Hudec M.D.<sup>1</sup>
Kamil Vrbica M.D.<sup>1</sup>
Jan Stasek M.D., EDIC<sup>1</sup>
Kateřina Rusinova M.D. MgA., Ph.D.<sup>2</sup>
prof. Andrea Pokorna PhDr., Ph.D.<sup>3</sup>
Jan Malaska M.D., Ph.D., EDIC<sup>1</sup>

## Affiliations:

- <sup>1)</sup> Department of Anesthesiology and Intensive Care Medicine, University Hospital Brno and Faculty of Medicine, Masaryk University, Brno, Czech Republic.
- <sup>2)</sup> Department of Anaesthesiology and Intensive Care, First Faculty of Medicine, Charles University in Prague and General University Hospital in Prague, Prague, Czech Republic <sup>3)</sup> Department of Health Sciences, Faculty of Medicine, Masaryk University, Brno, Czech Republic

Description: Pandemic of coronavirus SARS-CoV-2 (Severe Acute Respiratory Syndrome coronavirus 2) causing the disease COVID-19 (Coronavirus Disease 2019) overwhelmed healthcare and brought new challenges and stressful situations. In a short time, intensive care units (ICU) capacities were filled in many countries and regions. Due to the need for an excessive number of patients requiring intensive care, physicians and nurses who do not routinely provide care to critically ill patients or do not have the appropriate training (non-ICU clinician) were involved in the care of COVID-19 patients. In this context, ICU directly dedicated to caring for patients with COVID-19 ARDS (Acute Respiratory Distress Syndrome) was also opened. Non-ICU clinicians were more or less involved together with the standard ICU staff in palliative care, including End-of-Life decision (EOLD) making, even in a situation of limited, scarce resources (equipment or personnel). New workplace and scope of work, which did not correspond to the standard activity or education, most likely led to an increased stress load. EOLD can also be one of the factors leading to increased stress levels. The project aims to describe the practice of palliative care for patients with COVID-19 in a situation of pandemic COVID-19 and to identify factors leading to possible moral distress related to EOLD.

**Target group:** Healthcare providers (physicians and nurses) providing care to patients with COVID-19 admitted at ICU in the period of COVID-19 pandemic. (ICU – intensive care unit is defined in this study as a department with the possibility of mechanical ventilation)

**Primary outcome:** Description of the practice of providing palliative care, including EOLD practice in patients with COVID-19 admitted at ICU in COVID-19 pandemic.

## **Secondary outcome:**

a) Identify factors leading to moral distress during the COVID-19 pandemic

b) Describe possible different factors of moral distress by profession

**HO:** The process of providing palliative care, including End-of-life decisions, do not differ according to the type of workplace, demographic characteristics of healthcare providers, their education and job title. The level of moral distress in the situation of the COVID-19 pandemic in the period 2020/2021 was the same as before the pandemic. Factors associated with moral distress did not differ according to the communication, workplace safety, not even by job title.

Period of study: 1<sup>st</sup> July 2021 – 31<sup>st</sup> December 2021

Type of project: standard research

## Study design:

-Study type: observational descriptive non-interventional study

-Model of observational study: a survey study

-Time perspective: prospective -Biological material: none

-Number of groups/cohorts: 2 – (physicians and nurses)

**Randomisation:** Purposive sampling (Participants were included because they met inclusion criteria.

**Exclusion criteria:** Healthcare professionals who did not manage COVID-19 patients admitted at the ICU in the situation of COVID-19 pandemic in the period 2020/2021.

**Risks/BIAS:** Survey studies have their limitations, and the proposed survey is no exception. The risk is an insufficient research sample. The risk will be eliminated by choosing suitable research assistants and contact persons and cooperating with professional organisations. The use of professional contacts and web portals focused on the provision of intensive care.

**Ethics Committee:** An application has been submitted by the Ethics Committee, Faculty of Medicine, Masaryk University, Brno.